CLINICAL TRIAL: NCT03787758
Title: A Phase 1, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Determine the Safety, Tolerability, and Pharmacokinetics of SAGE-718 Oral Solution in Healthy Adults With an Open-label Cohort of Patients With Huntington's Disease
Brief Title: A Study to Evaluate Safety, Tolerability, and Pharmacokinetics of SAGE-718 Oral Solution in Patients With Huntington's Disease - Part B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 718-CLP-102 B
Record Dates: First submitted 2018-12-17; First posted 2018-12-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2022-01

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SAGE-718 (Experimental)
  Interventions: Drug: SAGE-718

INTERVENTIONS:
Drug: SAGE-718 — SAGE-718

SUMMARY:
This study is a phase 1, double-blind, placebo-controlled, multiple ascending dose study to determine the safety, tolerability, and pharmacokinetics of SAGE-718 oral solution in healthy adults (Part A) with an open-label cohort of patients with Huntington's disease (Part B)

DETAILED DESCRIPTION:
This posting addresses Part B

ELIGIBILITY:
Inclusion Criteria:

1. Subject is positive for mutant HTT (documented CAG repeats ≥ 40 units).
2. Subject has a body weight ≥50 kg and body mass index ≥18.0 and ≤30.0 kg/m2 at screening.

Exclusion Criteria:

1. Subject has any clinically significant abnormal finding on the physical exam at screening or admission.
2. Subject has a history or presence of a neurologic disease or condition (other than Huntington's disease), including but not limited to severe chorea, epilepsy, closed head trauma with clinically significant sequelae, or a prior seizure.
3. Subject has a family history of epilepsy.
4. Subject has a positive screening test for alcohol or drugs of abuse (including marijuana) at screening or admission.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with the Incidence of Adverse Events and Serious Adverse Events. | 21 Days
Percentage of participants with change from baseline in vital signs. | 21 Days
Change from baseline in electrocardiograms (ECGs) including PR interval, QT interval, QTc interval, QTcF, and rhythm abnormalities | 21 Days
Percentage of participants with change from baseline in clinical laboratory parameters. | 21 Days
Change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS). | 21 Days

SECONDARY OUTCOMES:
PK profile of SAGE-718 following administration of multiple doses of SAGE-718 Oral Solution as assessed by area under the curve [AUC]. | 17 Days
PK profile of SAGE-718 following administration of multiple doses of SAGE-718 Oral Solution as assessed by maximum observed concentration [Cmax]. | 17 Days
PK profile of SAGE-718 following administration of multiple doses of SAGE-718 Oral Solution as assessed by time of occurrence of Cmax [tmax]. | 17 Days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sage Investigational Site, Long Beach, California
  - Sage Investigational Site, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- [Derived] Koenig A, Lewis M, Wald J, Li S, Varoglu M, Dai J, Sankoh A, Paumier K, Doherty J, Quirk M. Dalzanemdor (SAGE-718), a novel, investigational N-methyl-D-aspartate receptor positive allosteric modulator: Safety, tolerability, and clinical pharmacology in randomized dose-finding studies in healthy participants and an open-label study in participants with Huntington's disease. Clin Transl Sci. 2024 Jul;17(7):e13852. doi: 10.1111/cts.13852. PMID 38988035